CLINICAL TRIAL: NCT07394634
Title: Evaluating the Efficacy of Autogenous Tooth Graft (ATG) Material in Socket Preservation: A Clinical and Radiographic Study.
Brief Title: Efficiency of Self Extracted Tooth Graft in Extraction Socket : A Clinical and Radiographic Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mahsa University (Other)
Responsible Party: Principal Investigator, Lim Poh Ling, Dr, Mahsa University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RMC/JANUARY/2025/EC07
Record Dates: First submitted 2026-01-23; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self Healing Group (No Intervention): Self healing in extraction socket
- Autogenous tooth graft (Experimental): Autogenous tooth grafting in extraction socket
  Interventions: Procedure: autogenous tooth graft

INTERVENTIONS:
Procedure: autogenous tooth graft — Extracted tooth will be grind and processed into bone graft . This bone graft material will grafted into the extraction socket
  Arms: Autogenous tooth graft

SUMMARY:
This is the clinical trial. The goal of this clinical trial is to test whether self extracted tooth graft (autogenous tooth graft ) able to preserved the extraction socket effectively. Our aim is to answer is there any difference in dimensional changes in extraction socket in clinically and radiographically Researchers will compare autogenous tooth graft with self-healing extraction socket in radiographic and clinical measurement.

Participant will be randomly allocated into 2 groups ( Test or controlled group) Test group will be autogenous tooth grafting post extraction. After removed any caries, calculus and any gilling material, the extracted tooth will be grind with grinder and processed using BONMAKER machine. (which the bone graft is washed with hydrogen peroxide, hydrogen chloride and alcohol isopropyl) and controlled group will be self healing group. Both group will withdraw 20cc blood for PRF ( Plasma rich fibrin) membrane and place into the socket and secured with suture. They will be reviewed post extraction 1 week ( to ensure there is no infection ) , 2 week ( for suture removal ) , 1 months ( For clinical measurement) , 3 months (For clinical and radiographic measurement) and 6 months (For radiographic measurement).

ELIGIBILITY:
Inclusion Criteria:

1. Age> or equal to 18 years old
2. Presence of adjacent teeth to the extraction site
3. Healthy ,or well controlled systemic disease
4. Lower and upper incisors, lower premolar/ first molar
5. Full mouth plaque score < 15%
6. Adequate space for a dental implant restoration *Patient with previous diagnosis of periodontitis will be required to have a successfully completed course of periodontal treatment before enrolment.

Exclusion Criteria:

1. Smokers and vapers
2. Acute infection or sinus tract in relation to the tooth that require extraction
3. Pregnant or lactating women
4. Patient received antibiotic for past 1 month
5. Loss of more than 50% buccal or lingual /palatal bone at the time of extraction
6. Patient on medication that altered bone metabolism or bone healing such as bisphosphonates, chemotherapeutic drugs or immunosuppressive agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Socket dimensional changes in autogenous tooth graft group and self healing group | 6 months
  Socket dimensional changes will be measure in clinical and radiographic measure Clinical measure: A stent will be made prior extraction and hole on the stent will be made to standardized measurement. Clinical measurement ( socket height) will be measure during post extraction, 1 month, 3 month and 6 month to observe the value of the resorption of the extraction socket . The discrepancy value is will be from ( 1month -baseline, 3month-baseline, 6month- baseline)
  Radiographic measure: CBCT will be taken post extraction 3 month and 6month. Socket width will be measure in 3mm below the socket and 5 mm below the socket. Other than that, mimic software will be used for the volumetric changes.

SECONDARY OUTCOMES:
Volumetric changes in autogenous tooth group and self healing group | 6 months
  In this , mimic software will be used for volumetric changes

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistrty, Jenjarum, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Elfana A, El-Kholy S, Saleh HA, Fawzy El-Sayed K. Alveolar ridge preservation using autogenous whole-tooth versus demineralized dentin grafts: A randomized controlled clinical trial. Clin Oral Implants Res. 2021 May;32(5):539-548. doi: 10.1111/clr.13722. Epub 2021 Mar 1. PMID 33565656

DOCUMENTS (1):
  • Informed Consent Form (2026-01-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT07394634/ICF_000.pdf